CLINICAL TRIAL: NCT04576585
Title: Appetite Lexicon Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Purdue University (Other)
Responsible Party: Principal Investigator, Richard Mattes, Distinguished Professor, Purdue University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2020-214
Record Dates: First submitted 2020-09-10; First posted 2020-10-06 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Appetitive Behavior
MeSH Terms: conditions — Appetitive Behavior

STUDY DESIGN:
Intervention Model Description: Investigators will randomly assign recruited participants to one of two groups. One group will receive training in the lexicon of appetite (Hunger, Fullness, Desire to Eat, and Prospective Consumption), and the other group will be trained in the basic tastes (Sweetness, Sourness, Bitterness, and Saltiness) as an attention control. All participants will participate in two preload trials with mixed meals before training and six paired preload trials after training. Trials will be held once per week. On another day of the trial week, participants will record their appetite during the waking hours of one day through an online survey. The total duration of participation will be in 9 weeks.
Who Masked: Participant
Masking Description: randomly assigned
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Appetite lexicon training group (Experimental): They will get appetite lexicon training in week three.
  Interventions: Behavioral: Lexicon training
- taste Lexicon training (Active Comparator): They will get taste lexicon training In week three.
  Interventions: Behavioral: Lexicon training

INTERVENTIONS:
Behavioral: Lexicon training — Participants will receive training on the lexicon of appetite on up to 3 days during the training week. This will entail reading written definitions, watching an instructional video, eating exercises and completing training exams demonstrating they understand the distinctions between appetitive terms (hunger, desire to eat, fullness, and prospective consumption). The training will require about 30 minutes to complete. To ensure the success of training, participants must verbally describe the definitions of the outcome sensations to a member of the research team and complete a written quiz with at least 90 % correct responses. Failure to satisfactorily convey understanding of the concepts will result in an offer to repeat the training 2 more times or be rejected from the study.

SUMMARY:
A fundamental limitation to the application of appetitive sensations is how they are measured. The most common approach relies on untrained individuals to self-report the sensations they experience under a given set of conditions. Investigators believe this is problematic because assumptions made about participant ratings are likely not valid. The proposed protocol will permit examination of whether training on appetite lexicon enhances the reliability of appetite ratings. Investigators also hypothesize that different preloads will induce different magnitudes of appetite sensations (hunger, fullness, desire to eat, and prospective consumption) depending on their energy density.

DETAILED DESCRIPTION:
A fundamental limitation to the application of appetitive sensations is how they are measured. The most common approach relies on untrained individuals to self-report the sensations they experience under a given set of conditions. Investigators believe this is problematic because assumptions made about participant ratings are likely not valid. Most commonly, participants are asked to rate their hunger, desire to eat, fullness, and prospective consumption. For example, researchers have demonstrated that hunger and fullness stem from different physiological processes (e.g., different gut-peptides and neurotransmitters) and serve different purposes (eating initiation (hunger), meal termination (fullness)) and, accordingly, expect participants to rate the two sensations independently. However, participants treat them as opposite poles on a common continuum. Additionally, in focus group analysis, consumers often use researcher-defined distinct terms interchangeably (hunger=desire to eat; fullness =lack of desire to eat). However, the distinction between these sensations is clinically important. Hunger and fullness do not always change reciprocally and equally in clinical conditions. Hunger can change without a shift in fullness, and the reverse has also been reported. Investigators believe reporting sensitivity, selectivity, and reliability can be improved by training participants on the terminology of appetitive sensations prior to testing, just as any bench researcher would calibrate their instruments before measurements. The proposed protocol will permit examination of whether training on appetite lexicon enhances the reliability of appetite ratings. Investigators also hypothesize that different preloads will induce different magnitudes of appetite sensations (hunger, fullness, desire to eat, and prospective consumption) depending on their energy density.

ELIGIBILITY:
Inclusion Criteria:

1. BMI 18-25 kg/m2.
2. Age 18-60 years.
3. Body weight fluctuation of <2.5kg in the past 3 months.
4. Fasting blood glucose below 6.1mmol/1 via capillary finger-stick blood sample using a SureStep glucometer (Lifescan, Milpitas, CA).
5. Regular eating pattern (i.e., reliable timing of eating events (±1 hour at least 5 days/wk - absolute pattern is less important than consistency.))
6. Willing to eat all test foods. Exclusion

Exclusion Criteria:

1. Having an acute disease.
2. Planning to initiate or terminate the use of medication known to affect appetite.
3. Diagnosed relevant chronic health conditions (e.g. diabetes, cardiovascular disease).
4. Allergies to eggs, peanuts, gluten, dairy, and carrots.
5. Age 61+ years

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2020-08-25 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
specificity of responses | start of study, day 1
  to measure if training in appetite descriptors leads to more specific responses in the appetite questionnaire.
specificity of responses | study completion, 9 weeks
  to measure if training in appetite descriptors leads to more specific responses in the appetite questionnaire.
test reliability | start of study, day 1
  measure if training in appetite descriptors will result in higher reliability in the appetite questionnaire.
test reliability | study completion, 9 weeks
  measure if training in appetite descriptors will result in higher reliability in the appetite questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Richard D Mattes, PhD, Principal Investigator — Purdue University
Locations (1):
- Purdue Univeristy, West Lafayette, Indiana, United States